CLINICAL TRIAL: NCT00115362
Title: Serotonin Effect in Non-Ulcer Dyspepsia
Brief Title: Serotonin Effect in Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SEREIN
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Dyspepsia
Keywords: functional dyspepsia;; Serotonin Uptake Inhibitors;; Antidepressive Agents.
MeSH Terms: conditions — Dyspepsia | interventions — Venlafaxine Hydrochloride

INTERVENTIONS:
Drug: venlafaxine

SUMMARY:
The purpose of this study is to investigate whether Efexor (venlafaxine) is effective in the treatment of functional dyspepsia.

DETAILED DESCRIPTION:
BACKGROUND: A good 60% of patients presenting with upper abdominal complaints have functional dyspepsia. Usually, acid-suppressive drugs are given as first-line therapy for upper gastrointestinal symptoms. However, results are often not satisfying and symptoms persist. Since many patients with functional gastrointestinal diseases are more anxious and depressed in comparison to healthy controls, several studies investigated the use of antidepressant agents in these patients. Although many studies were underpowered, promising results were obtained with tricyclic antidepressant and mianserin in patients with irritable bowel syndrome. There is still a need for a placebo controlled study with antidepressants in patients with functional dyspepsia.

OBJECTIVE: To investigate the effectiveness of venlafaxine, a selective serotonin and norepinephrine reuptake inhibitor, for treatment of patients with functional dyspepsia.

STUDY DESIGN: A randomized, double blind, placebo controlled trial.

STUDY POPULATION: Consecutive patients with persistent upper GI symptoms without abnormalities at upper gastrointestinal endoscopy.

PRIMARY ENDPOINTS: Upper gastrointestinal symptom absence after 6 weeks treatment.

SECONDARY ENDPOINTS:

* Anxiety and depression after venlafaxine treatment;
* Health related quality of life after venlafaxine treatment;
* The association between serotonin transporter protein and 5-HT receptor polymorphisms and efficacy of venlafaxine.

STUDY PROCEDURE: A venous blood sample will be collected in a 10ml EDTA-tube. Then, each subject will be randomized to treatment with Efexor XR (first and last two weeks 75 mg 1dd and from the third to the fifth week 75 mg 2dd) or identical placebos for 8 weeks. Before starting and after finishing treatment, patients will be asked to fill out a questionnaire on intensity of their gastrointestinal complaints, current quality of life and anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Persistent upper gastrointestinal symptoms;
* Absence of any serious organic cause of the complaints at previous upper gastrointestinal endoscopy (including gastric ulcer, carcinoma, oesophageal reflux disease, portal hypertension, hernia hiatus >2 cm or severe gastritis);
* Over 18 years of age;
* Written informed consent.

Exclusion Criteria:

* History of bipolar disorder;
* Contra-indication for venlafaxine;
* Current or planned pregnancy or lactation;
* Diagnosed alcoholism, anorexia nervosa or bulimia;
* Current or recent (within the last two weeks) use of a selective serotonin re-uptake inhibitor (SSRI) or MAO-inhibitor;
* Any other condition or circumstance that, in the opinion of the investigator or the physician, would compromise the subject's successful participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Upper gastrointestinal symptom absence after 6 weeks treatment.

SECONDARY OUTCOMES:
Anxiety and depression after venlafaxine treatment
Health related quality of life after venlafaxine treatment
The association between serotonin transporter protein and 5-HT receptor polymorphisms and efficacy of venlafaxine.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jansen, Professor MD, Study Director — Radboud University Nijmegen Medical Center
Locations (6):
- Netherlands (6):
  - Radboud University Nijmegen Medical Center, Nijmegen, P.O. Box 9101
  - Rijnstate Hospital, Arnhem
  - Slingeland Hospital, Doetinchem
  - Gelderse Vallei Hospital, Ede
  - Canisius-Wilhelmina Hospital, Nijmegen
  - Bernhoven hospital, Oss